CLINICAL TRIAL: NCT03649165
Title: A Phase I, Open-label, Single-center Relative Bioavailability and Food Effect Randomized Crossover Study of New Granule and Capsule Formulations of Selumetinib (AZD6244) in Healthy Male Subjects
Brief Title: A Study to Evaluate Bioavailability and Food Effect of Selumetinib (AZD6244) in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D1532C00089
Record Dates: First submitted 2018-08-24; First posted 2018-08-28 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2018-11

CONDITIONS: Neurofibromatosis Type 1 (NF1)-Related Plexiform Neurofibromas (PNs); Healthy Participants
Keywords: MEK Inhibitor; Selumetinib capsule; Selumetinib granule; PK; Bioavailibilty; Crossover study; Open-label; Food effect
MeSH Terms: conditions — Neurofibromatosis 1 | interventions — Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment Sequence 1 (Experimental): Participants will receive Treatment A (selumetinib 25 mg granule, fasted state) in Part 1, Period 1, Treatment B (selumetinib 50 mg capsule, fasted state) in Part 1, Period 2, Treatment C (selumetinib 25 mg granule, fed state) in Part 2, Period 3, and Treatment D (selumetinib 50 mg capsule, fed state) in Part 2, Period 4. Participants will also receive a single 500 mg dose of acetaminophen at the same time as selumetinib administration where it will act as a marker for gastric emptying.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C; Drug: Treatment D; Drug: Acetaminophen
- Treatment Sequence 2 (Experimental): Participants will receive Treatment B (selumetinib 50 mg capsule, fasted state) in Part 1, Period 1, Treatment A (selumetinib 25 mg granule, fasted state) in Part 1, Period 2, Treatment C (selumetinib 25 mg granule, fed state) in Part 2, Period 3 and Treatment D (selumetinib 50 mg capsule, fed state) in Part 2, Period 4. Participants will also receive a single 500 mg dose of acetaminophen at the same time as selumetinib administration where it will act as a marker for gastric emptying.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C; Drug: Treatment D; Drug: Acetaminophen
- Treatment Sequence 3 (Experimental): Participants will receive Treatment A (selumetinib 25 mg granule, fasted state) in Part 1, Period 1, Treatment B (selumetinib 50 mg capsule, fasted state) in Part 1, Period 2, Treatment D (selumetinib 50 mg capsule, fed state) in Part 2, Period 3 and Treatment C (selumetinib 25 mg granule, fed state) in Part 2, Period 4. Participants will also receive a single 500 mg dose of acetaminophen at the same time as selumetinib administration where it will act as a marker for gastric emptying.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C; Drug: Treatment D; Drug: Acetaminophen
- Treatment Sequence 4 (Experimental): Participants will receive Treatment B (selumetinib 50 mg capsule, fasted state) in Part 1, Period 1, Treatment A (selumetinib 25 mg granule, fasted state) in Part 1, Period 2, Treatment D (selumetinib 50 mg capsule, fed state) in Part 2, Period 3 and Treatment C (selumetinib 25 mg granule, fed state) in Part 2, Period 4. Participants will also receive a single 500 mg dose of acetaminophen at the same time as selumetinib administration where it will act as a marker for gastric emptying.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C; Drug: Treatment D; Drug: Acetaminophen

INTERVENTIONS:
Drug: Treatment A — During Part 1 of the study, participants will receive single doses of selumetinib 25 mg granule under fasted conditions. The dose will be administered after an overnight fast of at least 10 hours. The IMP will be administered with approximately 240 mL of water. No food will be allowed for at least 4 hours post-dose.
Drug: Treatment B — During Part 1 of the study, participants will receive single doses of selumetinib 50 mg capsule under fasted conditions. The dose will be administered after an overnight fast of at least 10 hours. The IMP will be administered with approximately 240 mL of water. No food will be allowed for at least 4 hours post-dose.
Drug: Treatment C — During Part 2 of the study, participants will receive single doses of selumetinib 25 mg granule under fed conditions. Following an overnight fast of at least 10 hours, participants will start consumption of the recommended meal within 30 minutes before administration of the IMP. Participants will be required to consume the entire meal in 30 minutes or less; however, the IMP should be administered 30 minutes after start of the meal. The IMP will be administered with approximately 240 mL of water. No food will be allowed for at least 4 hours post-dose, where after a meal may be provided.
Drug: Treatment D — During Part 2 of the study, participants will receive single doses of selumetinib 50 mg capsule under fed conditions. Following an overnight fast of at least 10 hours, participants will start consumption of the recommended meal within 30 minutes before administration of the IMP. Participants will be required to consume the entire meal in 30 minutes or less; however, the IMP should be administered 30 minutes after start of the meal. The IMP will be administered with approximately 240 mL of water. No food will be allowed for at least 4 hours post-dose, where after a meal may be provided.
Drug: Acetaminophen — Participants will receive a single 500mg dose of acetaminophen at the same time.

SUMMARY:
This study will evaluate bioavailability and food effect of selumetinib (AZD6244) in healthy male participants. A total of 24 healthy male participants will be included to ensure at least 20 evaluable participants. The study is divided in 2 study parts; the same participants will participate in both parts of the study. Part 1 of the study is to investigate the pharmacokinetics (PK) of the selumetinib granule compared to the PK of selumetinib capsule, when administered with water under the fasted conditions. Part 2 of the study is to investigate the PK of selumetinib granule and capsule under fed conditions. Participants will also receive a single 500 mg dose of acetaminophen at the same time as selumetinib administration.

DETAILED DESCRIPTION:
This study will be a 2-part, open-label, single-center relative bioavailability and food effect randomized crossover study of new granule and capsule formulations of selumetinib. A total of 24 healthy male participants aged between 18 to 45 years (inclusive), will be included to ensure at least 20 evaluable participants. The study is divided in 2 study parts; the same participants will participate in both parts of the study.

Part 1 of the study is designed to investigate the PK of the selumetinib granule compared to the PK of selumetinib capsule, when administered with water under the fasted conditions. Part 2 of the study is designed to investigate the PK of selumetinib granule and capsule under fed conditions. Participants will consume a low-fat, low-calorie meal. Thirty minutes after the start of the meal, selumetinib will be administered to the participants. In all treatment periods, participants will also receive a single 500 mg dose of acetaminophen at the same time as selumetinib administration where it will act as a marker for gastric emptying. The study will also assess the palatability of the selumetinib granule in both parts of the study.

Each participant will receive the following treatments:

* Treatment A: 25 mg granule, fasted state
* Treatment B: 50 mg capsule, fasted state
* Treatment C: 25 mg granule, fed state
* Treatment D: 50 mg capsule, fed state Participant will be randomly assigned to 1 of 4 treatment sequences. In all cases the treatments in Part 1 will be administered before the treatments in Part 2. The study will comprise of a screening period of maximum 28 days. Four treatment periods during which participants will be resident from the day before dosing (Day -1) until at least 48 hours after dosing; discharged on the morning of Day 3. A follow-up visit, will be within 7 to 10 days after the last dose of investigational medicinal product (IMP). There will be a minimum washout period of at least 5 days between each IMP administration. Each participant will be involved in the study for approximately 8 to 9 weeks.

ELIGIBILITY:
Inclusion Criteria

1. Provision of signed and dated, written informed consent before any study-specific procedures.
2. Healthy male participants aged 18 to 45 years (inclusive) with suitable veins for cannulation or repeated venipuncture.
3. Have a body mass index (BMI) between 18 and 30 kg/m2 inclusive and weigh at least 50 kg.
4. Participants is able to consume a low-fat meal within a 30-minute period.
5. Participants has a creatinine clearance (CRCL) greater than 50 mL/min using Cockcroft-Gault formula.
6. Participants is willing to comply with contraception requirements as described below:

   * Male participants with sexual partners who can become pregnant (i.e., women of childbearing potential) must use 2 highly-effective methods of contraception, one of which must be a barrier method (condom with spermicide) from the time of the first administration of the IMP until 12 weeks after the last administration of the IMP to avoid pregnancy and/or potential adverse effects on the developing embryo.
   * Participants with sexual partners who are pregnant must use an effective method of contraception (barrier method) from the time of the first administration of the IMP until 12 weeks after the last administration of the IMP.
   * Participants must avoid sperm donation during the study and for 12 weeks after the last administration of the IMP.
   * Reliable methods of contraception must be used consistently and correctly.
   * Reliable methods of contraception for participants include: Use of barrier methods (condom and spermicide) for the duration of the study until 12 weeks after the last administration of the IMP.
   * Acceptable methods for participants partners include:

     1. Use of implants, injectables and combined oral contraceptives (must be used in combination with a barrier method of contraception)
     2. Use of intrauterine devices (must be used in combination with a barrier method of contraception)

Exclusion Criteria :

1. Participants of Japanese, non-Japanese Asian or Indian ethnicity.
2. Participants has any one parent or grandparent (maternal or paternal) that was Japanese or non-Japanese Asian (e.g., China, Taiwan, Korea, Philippines, Thailand, Vietnam and Malaysia) or Indian.
3. History or presence of central serous retinopathy or retinal vein thrombosis, IOP greater than 21 mmHg or uncontrolled glaucoma.
4. History of any clinically significant disease or disorder which, in the opinion of the PI, may put the participant at risk because of participation in the study, influence the result of the study or influence the participants ability to participate in the study.
5. Participant has ophthalmologic conditions as follows:

   * Current or past history of central serous retinopathy/retinal pigment epithelial detachment or retinal vein occlusion.
   * Intra-ocular pressure > 21 mmHg or uncontrolled glaucoma (irrespective of IOP).
6. Participant has any cardiac conditions as follows:

   * Uncontrolled hypertension (BP ≥ 150/95 mmHg despite medical therapy).
   * Acute coronary syndrome within 6 months before starting treatment.
   * Uncontrolled Angina - Canadian Cardiovascular Society grade II-IV despite medical therapy.
   * Symptomatic heart failure New York Heart Association (NYHA) Class II-IV, prior or current cardiomyopathy, or severe valvular heart disease.
   * Prior or current cardiomyopathy including but not limited to the following: 1) Known hypertrophic cardiomyopathy.

     2) Known arrhythmogenic right ventricular cardiomyopathy. 3) Previous moderate or severe impairment of LVEF < 45% on echocardiography even if full recovery has occurred.
   * Left ventricular ejection fraction below the lower limit of normal (LLN) or < 55% measured by ECHO at the Screening Visit.
   * Severe valvular heart disease.
   * Atrial fibrillation with a ventricular rate > 100 beats per minute (bpm) on ECG at rest.
   * QTcF > 450 ms or other factors that increase the risk of QT prolongation.
7. Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of IMP.
8. Any clinically relevant abnormal findings in physical examination, hematology, clinical chemistry, urinalysis, vital signs or ECG at the Screening Visit, which in the opinion of the PI, may put the participant at risk because of his participation in the study. Test may be repeated twice at the discretion of the Investigator if abnormal.
9. Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody, and human immunodeficiency virus (HIV) antibody.
10. A suspected/manifested infection according to the International Air Transport Association (IATA) Categories A and B infectious substances.
11. History of, or current alcohol or drug abuse, as judged by the principal investigator (PI).
12. Participation in another clinical study (investigational product administered within 30 days before the Screening Visit, or participation in a method development study [no drug] 30 days before the Screening Visit). Participation is defined as the completion of a treatment related visit.
13. Planned in-patient surgery, dental procedure or hospitalization during the study.
14. Plasma donation within 30 days of the Screening Visit or any blood donation/loss more than 500 mL during the 90 days before the Screening Visit.
15. A definite or suspected personal history of intolerance or hypersensitivity to drugs and/or their excipients, judged to be clinically relevant by the PI.
16. Known severe hypersensitivity to selumetinib or acetaminophen or any excipient of these medicinal products or history of allergic reactions attributed to compounds of similar chemical or biologic composition to selumetinib.
17. Current smokers or those who have smoked or used nicotine products (including e-cigarettes) within the 90 days before the Screening Visit.
18. Positive screen for drugs of abuse, alcohol or cotinine at the Screening Visit or on each admission to the Clinical Unit or positive screen for alcohol on each admission to the Clinical Unit.
19. Use of drugs with enzyme-inducing properties such as St John's Wort within 4 weeks before the first administration of IMP.
20. Use of any prescribed medicine and over-the-counter (OTC) drugs (including herbal remedies, vitamins and minerals) within 2 weeks or 5 times the half-life, whichever is the longer, of the respective drug before Day -1 or Treatment Period 1. No medications known to prolong the QT/QTc interval are allowed.
21. Excessive intake of caffeine-containing drinks or food e.g., coffee, tea, chocolate, Red Bull or cola (more than 6 units of caffeine per day). One caffeine unit is contained in the following items: 1 (6 oz) cup of coffee, 2 (12 oz) cans of cola, 1 (12 oz) cup of tea, ½ (4 oz) cup of energy drink (e.g., Red Bull) or 3 oz of chocolate.
22. Known or suspected history of alcohol or drug abuse or excessive intake of alcohol as judged by the PI.
23. Involvement of any AstraZeneca, PAREXEL or Clinical Unit employee or their close relatives.
24. Participants who have previously been randomized to treatment in the current study.
25. Judgment by the PI that the participant should not participate in the study if they have any ongoing or recent (i.e., during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions and requirements.
26. Vulnerable participants , e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 24 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2018-10-21 (Actual); Study Completion 2018-10-21 (Actual)

PRIMARY OUTCOMES:
Selumetinib and N-desmethyl selumetinib plasma PK parameter: Dose normalized area under plasma concentration-time curve from time zero to infinity (AUC/D) | At pre-dose, and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36 and 48 hours post-dose(Days -1 to 3)
  To compare the AUC/D of the new selumetinib granule formulation with selumetinib capsule formulation in fasted state.
Selumetinib and N-desmethyl selumetinib plasma PK parameter: Dose normalized area under the plasma concentration-time curve from time zero to time of last quantifiable concentration (AUClast/D) | At pre-dose, and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36 and 48 hours post-dose(Days -1 to 3)
  To compare the AUClast/D of the new selumetinib granule formulation with selumetinib capsule formulation in fasted state.
Selumetinib and N-desmethyl selumetinib plasma PK parameter: Dose normalized maximum observed plasma concentration (Cmax/D) | At pre-dose, and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36 and 48 hours post-dose(Days -1 to 3)
  To compare the Cmax/D of the new selumetinib granule formulation with selumetinib capsule formulation in fasted state.
Selumetinib and N-desmethyl selumetinib plasma PK parameter: Fraction of administered selumetinib granule dose systemically available relative to the capsule reference (Frel) | At pre-dose, and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36 and 48 hours post-dose(Days -1 to 3)
  To compare the Frel. of the new selumetinib granule formulation with selumetinib capsule formulation in fasted state.

SECONDARY OUTCOMES:
Selumetinib and N-desmethyl selumetinib plasma PK parameter: Area under plasma concentration time curve from time zero to infinity (AUC) | At pre-dose, and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36 and 48 hours post-dose(Days -1 to 3)
  To compare AUC of selumetinib capsule fasted versus capsule low-fat fed state.
Selumetinib and N-desmethyl selumetinib plasma PK parameter: Area under the plasma concentration time curve from time zero to time of last quantifiable concentration (AUClast) | At pre-dose, and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36 and 48 hours post-dose (Days -1 to 3)
  To compare AUClast of selumetinib capsule fasted versus capsule low-fat fed state.
Selumetinib and N-desmethyl selumetinib plasma PK parameter: Area under the plasma concentration-time curve from zero to 12 hours post-dose [AUC(0-12)] | At pre-dose, and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36 and 48 hours post-dose (Days -1 to 3)
  To compare AUC (0-12) of selumetinib capsule fasted versus capsule low-fat fed state.
Selumetinib and N-desmethyl selumetinib plasma PK parameter: Maximum observed plasma concentration (Cmax) | At pre-dose, and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36 and 48 hours post-dose (Days -1 to 3)
  To compare Cmax of selumetinib capsule fasted versus capsule low-fat fed state.
Selumetinib and N-desmethyl selumetinib plasma PK parameter: Ratio of AUC in fed state to AUC in the fasted state (FRAUC) | At pre-dose, and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36 and 48 hours post-dose (Days -1 to 3)
  To compare FRAUC of selumetinib capsule fasted versus capsule low-fat fed state.
Selumetinib and N-desmethyl selumetinib plasma PK parameter: Ratio of Cmax in fed state to Cmax in the fasted state (FRCmax) | At pre-dose, and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36 and 48 hours post-dose (Days -1 to 3)
  To compare FRCmax of selumetinib capsule fasted versus capsule low-fat fed state.
Selumetinib and N-desmethyl selumetinib plasma PK parameter: Half-life associated with terminal slope (λz) of a semi-logarithmic concentration-time curve (t½λz) | At pre-dose, and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36 and 48 hours post-dose (Days -1 to 3)
  To compare t½λz of selumetinib capsule fasted versus capsule low-fat fed state.
Selumetinib and N-desmethyl selumetinib plasma PK parameter: Time to reach maximum observed plasma concentration (tmax) | At pre-dose, and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36 and 48 hours post-dose (Days -1 to 3)
  To compare tmax of selumetinib capsule fasted versus capsule low-fat fed state.
Selumetinib and N-desmethyl selumetinib plasma PK parameter: Terminal elimination rate constant (λz) | At pre-dose, and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36 and 48 hours post-dose (Days -1 to 3)
  To compare λz of selumetinib capsule fasted versus capsule low-fat fed state.
Selumetinib plasma PK parameters: Apparent total body clearance of drug from plasma after extravascular administration (parent drug only) (CL/F) | At pre-dose, and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36 and 48 hours post-dose (Days -1 to 3)
  To compare CL/F of selumetinib capsule fasted versus capsule low-fat fed state.
Selumetinib plasma PK parameters: Apparent volume of distribution during the terminal phase after extravascular administration (Vz/F) | At pre-dose, and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36 and 48 hours post-dose (Days -1 to 3)
  To compare Vz/F of selumetinib capsule fasted versus capsule low-fat fed state.
Selumetinib and N-desmethyl selumetinib plasma PK parameter: AUC | At pre-dose, and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36 and 48 hours post-dose (Days -1 to 3)
  To compare AUC of selumetinib granule fasted versus granule low-fat fed state.
Selumetinib and N-desmethyl selumetinib plasma PK parameter: AUClast | At pre-dose, and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36 and 48 hours post-dose (Days -1 to 3)
  To compare AUClast of selumetinib granule fasted versus granule low-fat fed state.
Selumetinib and N-desmethyl selumetinib plasma PK parameter: AUC(0-12) | At pre-dose, and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36 and 48 hours post-dose (Days -1 to 3)
  To compare AUC (0-12) of selumetinib granule fasted versus granule low-fat fed state.
Selumetinib and N-desmethyl selumetinib plasma PK parameter: Cmax | At pre-dose, and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36 and 48 hours post-dose (Days -1 to 3)
  To compare Cmax of selumetinib granule fasted versus granule low-fat fed state.
Selumetinib and N-desmethyl selumetinib plasma PK parameter: FRAUC | At pre-dose, and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36 and 48 hours post-dose (Days -1 to 3)
  To compare FRAUC of selumetinib granule fasted versus granule low-fat fed state.
Selumetinib and N-desmethyl selumetinib plasma PK parameter: FRCmax | At pre-dose, and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36 and 48 hours post-dose (Days -1 to 3)
  To compare FRCmax of selumetinib granule fasted versus granule low-fat fed state.
Selumetinib and N-desmethyl selumetinib plasma PK parameter: t½λz | At pre-dose, and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36 and 48 hours post-dose (Days -1 to 3)
  To compare t½λz of selumetinib granule fasted versus granule low-fat fed state.
Selumetinib and N-desmethyl selumetinib plasma PK parameter: tmax | At pre-dose, and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36 and 48 hours post-dose (Days -1 to 3)
  To compare tmax of selumetinib granule fasted versus granule low-fat fed state.
Selumetinib and N-desmethyl selumetinib plasma PK parameter: λz | At pre-dose, and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36 and 48 hours post-dose (Days -1 to 3)
  To compare λz of selumetinib granule fasted versus granule low-fat fed state.
Selumetinib plasma PK parameters: CL/F | At pre-dose, and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36 and 48 hours post-dose (Days -1 to 3)
  To compare CL/F of selumetinib granule fasted versus granule low-fat fed state.
Selumetinib plasma PK parameters: Vz/F | At pre-dose, and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36 and 48 hours post-dose (Days -1 to 3)
  To compare Vz/F of selumetinib granule fasted versus granule low-fat fed state.
Taste questionnaire | At Days -1 to 3 (within 10 minutes following intake of selumetinib granule)
  To assess palatability of selumetinib granule formulation. The standardized questionnaire will be administered to participants within 10 minutes following intake of selumetinib granule. Questionnaire about taste include sweet, salty, sour, bitter, metallic, and hot/spicy. Where 0 indicates not at all and 10 indicates extremely.
Number of participants with adverse events (AEs) | From the time of informed consent, throughout the treatment periods up to and including the Follow-up Visit (7 to 10 days after last dose)
  To assess the safety and tolerability of single doses of selumetinib in healthy participants.
Vital signs (systolic blood pressure [BP]) | Change from baseline up to follow-up/early termination visit (7 to 10 days after last dose)
  To assess systolic BP as a variable of safety and tolerability of single doses of selumetinib in healthy participants. Participants should be supine and at rest for at least 5 minutes before the measurements.
Vital signs (diastolic BP) | Change from baseline up to follow-up/early termination visit (7 to 10 days after last dose)
  To assess diastolic BP as a variable of safety and tolerability of single doses of selumetinib in healthy participants. Participants should be supine and at rest for at least 5 minutes before the measurements.
Pulse rate | Change from baseline up to follow-up/early termination visit (7 to 10 days after last dose)
  To assess pulse rate as a variable of safety and tolerability of single doses of selumetinib in healthy participants.
  Participants should be supine and at rest for at least 5 minutes before the measurements.
12-lead electrocardiogram (ECG) | From baseline up to follow-up/early termination visit (7 to 10 days after last dose)
  To assess 12-lead ECG as variable of safety and tolerability of single doses of selumetinib in healthy participants. Participants should be supine and at rest 10 minutes before recording the ECG.
Number of participants with abnormal findings in physical examination | From baseline up to follow-up/early termination visit (7 to 10 days after last dose)
  To assess physical examination as a variable safety and tolerability of single doses of selumetinib in healthy participants.
Ophthalmic examinations | At screening Visit or on Day -1 of Treatment Period 1
  To assess ophthalmic examination as a variable of safety and tolerability of single doses of selumetinib in healthy participants. Ophthalmic examination included best corrected visual acuity, intra-ocular pressure and slit-lamp fundoscopy.
Laboratory assessments: hematology - Hemoglobin (Hb) | Change from baseline up to follow-up/early termination visit (7 to 10 days after last dose)
  To assess Hb as a variable of safety and tolerability of single doses of selumetinib in healthy participants.
Laboratory assessments: hematology - erythrocyte count | Change from baseline up to follow-up/early termination visit (7 to 10 days after last dose)
  To assess erythrocyte count as a variable of safety and tolerability of single doses of selumetinib in healthy participants.
Laboratory assessments: hematology: Platelet count | Change from baseline up to follow-up/early termination visit (7 to 10 days after last dose)
  To assess platelet count as a variable of safety and tolerability of single doses of selumetinib in healthy participants.
Laboratory assessments: hematology: leucocyte differential count (absolute count) | Change from baseline up to follow-up/early termination visit (7 to 10 days after last dose)
  To assess leucocyte differential count as a variable of safety and tolerability of single doses of selumetinib in healthy participants.
Laboratory assessments: hematology: leucocyte cell count | Change from baseline up to follow-up/early termination visit (7 to 10 days after last dose)
  To assess leucocyte cell count as variable of safety and tolerability of single doses of selumetinib in healthy participants.
Laboratory assessments:hematology - differential count | Change from baseline up to follow-up/early termination visit (7 to 10 days after last dose)
  To assess differential count of neutrophils, lymphocytes, monocyets, eosinophils and basophils) as a variable of safety and tolerability of single doses of selumetinib in healthy participants.
Laboratory assessments: Serum clinical chemistry - electrolytes | Change from baseline up to follow-up/early termination visit (7 to 10 days after last dose)
  To assess serum level of sodium, potassium, magnesium and phosphate as a variable of safety and tolerability of single doses of selumetinib in healthy participants.
Laboratory assessments: Serum clinical chemistry - urea nitrogen | Change from baseline up to follow-up/early termination visit (7 to 10 days after last dose)
  To assess urea nitrogen as a variable of safety and tolerability of single doses of selumetinib in healthy participants.
Laboratory assessments: Serum clinical chemistry - creatinine | Change from baseline up to follow-up/early termination visit (7 to 10 days after last dose)
  To assess creatinine as variable of safety and tolerability of single doses of selumetinib in healthy participants.
Laboratory assessments: Serum clinical chemistry: albumin | Change from baseline up to follow-up/early termination visit (7 to 10 days after last dose)
  To assess albumin as a variable of safety and tolerability of single doses of selumetinib in healthy participants.
Laboratory assessments: Serum clinical chemistry: Total Calcium | Change from baseline up to follow-up/early termination visit (7 to 10 days after last dose)
  To assess total calcium as a variable of safety and tolerability of single doses of selumetinib in healthy participants.
Laboratory assessments: Serum clinical chemistry: Total protein | Change from baseline up to follow-up/early termination visit (7 to 10 days after last dose)
  To assess total protein as a variable of safety and tolerability of single doses of selumetinib in healthy participants.
Laboratory assessments: Serum clinical chemistry: Total bilirubin | Change from baseline up to follow-up/early termination visit (7 to 10 days after last dose)
  To assess total bilirubin as a variable of safety and tolerability of single doses of selumetinib in healthy participants.
Laboratory assessments: Serum clinical chemistry: Creatine phosphokinase (CPK) | Change from baseline up to follow-up/early termination visit (7 to 10 days after last dose)
  To assess CPK as a variable of safety and tolerability of single doses of selumetinib in healthy participants.
Laboratory assessments: Serum clinical chemistry: Troponin (isoform as per institutional norm) | Change from baseline up to follow-up/early termination visit (7 to 10 days after last dose)
  To assess troponin as a variable of safety and tolerability of single doses of selumetinib in healthy participants.
Laboratory assessments: Serum clinical chemistry - Liver enzymes | Change from baseline up to follow-up/early termination visit (7 to 10 days after last dose)
  To assess serum of Alkaline phosphatase (ALP), Alanine aminotransferase (ALT), Aspartate aminotransferase (AST) and Gamma glutamyl transpeptidase (GGT) as a variable of safety and tolerability of single doses of selumetinib in healthy participants.
Laboratory assessments: Clinical urinalysis - glucose | Change from baseline up to follow-up/early termination visit (7 to 10 days after last dose)
  To assess urine glucose as a variable of safety and tolerability of single doses of selumetinib in healthy participants.
Laboratory assessments: Clinical Urinalysis - protein | Change from baseline up to follow-up/early termination visit (7 to 10 days after last dose)
  To assess urine protein as a variable of safety and tolerability of single doses of selumetinib in healthy participants.
Laboratory assessments: Clinical Urinalysis - blood | Change from baseline up to follow-up/early termination visit (7 to 10 days after last dose)
  To assess urine blood as a variable of safety and tolerability of single doses of selumetinib in healthy participants.
  If urinalysis is positive for blood, a microscopy test will be performed to assess RBC, white blood cell [WBC], casts [cellular, granular, hyaline]).

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Goldwater, MD, Principal Investigator — PAREXEL Early Phase Clinical Unit Baltimore
Locations (1):
- Research Site, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cohen-Rabbie S, Mattinson A, So K, Wang N, Goldwater R. A Phase I, Open-label, Randomized, Crossover Study of the Relative Bioavailability of Capsule and Granule Formulations of Selumetinib. Clin Ther. 2022 Apr;44(4):565-576. doi: 10.1016/j.clinthera.2022.02.009. Epub 2022 Apr 9. PMID 35410754
- [Derived] Cohen-Rabbie S, Mattinson A, So K, Wang N, Goldwater R. Effect of food on capsule and granule formulations of selumetinib. Clin Transl Sci. 2022 Apr;15(4):878-888. doi: 10.1111/cts.13209. Epub 2022 Feb 15. PMID 35170228